CLINICAL TRIAL: NCT05743608
Title: Non-interventional, Open-label, Prospective Study to Assess the Effectiveness of BDP/FF/G Fixed Triple Inhalation Powder on Symptom Scores in Moderate to Severe COPD Patients, Uncontrolled With Inhaled Dual Therapies (LABA/LAMA or ICS/LABA)
Brief Title: NEXThaleR Real-world Study Assessing the EffectivenesS of BDP/FF/G Fixed triPle cOmbiNation on Symptom scorEs in COPD Patients
Acronym: RESPONSE
Status: Completed | Type: Observational
Sponsor: Chiesi Hungary Ltd. (Industry)
Collaborators: Chiesi Slovenija, d.o.o. (Industry); Chiesi Bulgaria (Industry); CHIESI CZ s.r.o. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHMED_2022/01
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: COPD; CAT; Fixed-dose triple inhaled therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to severe COPD patients receiving Trimbow dry powder inhaler: Patients above the age of 35 years, who had been diagnosed with COPD for over a year by a pulmonologists specialist. Having a moderate or severe obstruction (30%≤FEV1<80%) and are uncontrolled despite fixed dual combination treatment (LABA/LAMA or ICS/LABA). Therapy was changed to Trimbow® 88/5/9 µg inhalation powder maximum 1 week prior to or on the day of study inclusion and irrespective of study entry (escalation of symptomatic patient to fixed triple combination as per treatment protocol)

SUMMARY:
The goal of this observational study is to measure improvement in health related quality of life in moderate to severe COPD patients treated with Trimbow inhalation powder. The main question[s] it aims to answer are:

* Treatment's effect on quality of life
* Treatment's effect on lung function Participants will be assessed according to routine clinica practice, without any additional intervention.

DETAILED DESCRIPTION:
COPD is a severe and very common disease affecting a large proportion of smokers (and even non-smokers) all around the world. With the large prevalence and wide spectrum of disease presentation (from limited obstruction to life threatening conditions) there is a need for differentiated, targeted approach to therapy. For this purpose, plenty of inhaler devices had been developed. Chiesi is the only company which provides fix triple combinations in both DPI and pMDI formulations. While there is ample data from multiple studies on the real-world effectiveness of the pMDI, there is a relevant gap in our knowledge on the RWE effectiveness of the DPI device Trimbow dry powder inhaler is a novel extrafine, single inhaler triple therapy, in a state of the art dry powder inhaler, which is easy to use and may provide additional benefit to a large proportion of COPD patients. However, there are only a limited number of studies assessing its effectiveness, especially in patients with moderate airflow obstruction. Providing more real-world evidence that Trimbow® dry powder inhaler is an effective and preferred treatment option in reducing symptoms and improving lung function in all COPD patients, would help pulmonologists choose the most suitable treatment option for a very wide array of patients.

ELIGIBILITY:
Inclusion criteria:

* Patient had been diagnosed with COPD for over a year by a pulmonologists specialist
* Patients ≥ 35 years of age
* outpatient
* Having had a spirometry test performed maximum 1 month prior to inclusion OR on the day of study inclusion
* Eligibility to Trimbow 88/5/9 µg inhalation powder treatment according to SmPC:

  * having a moderate or severe obstruction (30%≤FEV1<80%)
  * uncontrolled despite fixed dual combination treatment (LABA/LAMA or ICS/LABA):

    * at least 1 severe or 2 moderate exacerbations (requiring hospital admission) in the past 12 months
    * symptomatic patient (CAT≥10 and/or mMRC ≥2)
* Therapy was changed to Trimbow® 88/5/9 µg inhalation powder maximum 1 week prior to or on the day of study inclusion and irrespective of study entry (escalation of symptomatic patient to fixed triple combination as per treatment protocol)
* Patient provided informed consent to study participation and related data collected
* Patient with no functional disability

Exclusion criteria:

* Participation in any clinical trial, 30 days prior to inclusion
* Ongoing severe exacerbation (requiring hospitalisation) or severe exacerbation within the last 4 weeks
* Diagnosis of asthma (asthma/COPD co-occurrence - ACO not allowed!)
* Continuous use of oral corticosteroids or oxygen therapy
* Patients with other important diseases of the respiratory system or other organ systems that may significantly contribute to COPD symptoms (such as untreated heart failure, symptomatic anaemia, etc.)
* Any additional contraindications listed in the SmPC for Trimbow® 88/5/9 µg inhalation powder and any other provision in the SmPC that would prevent the patient from receiving fixed triple combination therapy
* The patient is unable to complete the part of the questionnaire(s) relevant to him/her

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe COPD patients who are uncontrolled on either LABA/LAMA or ICS/LABA fixed dose dual combination therapy, and had been switched to Trimbow dry powder inhaler prior to study inclusion
Sampling Method: Non-Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 6 months
  Change in symptom scores (COPD Assessment Test - CAT) after six months of treatment. On a scale of 0-40

SECONDARY OUTCOMES:
Lung function - Forces Expiratory flow in 1 second (FEV1) | 6 months
  Change in FEV1 values after inhalation during 6 months of treatment compared to baseline.
Lung function Forced Vital Capacity (FVC) | 6 months
  Change in FVC values after inhalation during 6 months of treatment compared to baseline.
Responders | 6 months
  Percentage of patients with a change from baseline 2< in CAT after 6 months of treatment compared to baseline (assessment of response to therapy).
Health Related Quality of Life (HRQoL) - questions | 6 months
  To assess changes in quality of life in EQ-5D-3L domains after 6 months of treatment compared to baseline. Scale on a level of three
HRQoL - VAS | 6 months
  To assess changes in quality of life in EQ-5D visual analogue scale (VAS) after 6 months of treatment compared to baseline. Scale from 0-100
Symptoms | 6 months
  To assess changes in frequency of cough and sputum production after 6 months of treatment compared to baseline.
Saturation | 6 months
  To assess changes in arterial oxygenation compared to baseline oxigen saturation (SpO2) after 6 months of treatment.
Adherence | 6 months
  To assess changes in adherence to inhaler treatment according to the TAI (Test of adherence to inhalers) questionnaire after 6 months of treatment compared to baseline. Scale is from 12-54
Night-time symptoms | 6 months
  To assess changes in the frequency of night-time symptoms after 6 months of treatment compared to baseline.
mMRC | 6 months
  To assess changes in dyspnoea severity using the mMRC (modified Medical Research Council) questionnaire after 6 months of treatment compared to baseline. Scale from 1-4

CONTACTS AND LOCATIONS:
Locations (39):
- Hungary (39):
  - Albert Schweitzer Kórház és Rendelőintézet Tüdőbeteggondozó, Aszód
  - Bajai Szent Rókus Kórház, Tüdőbeteggondozó Intézet, Baja
  - National Korányi Institute of Pulmonology, Budapest
  - Bajcsy -Zsilinszky Kórház és Rendelőintézet, Budapest
  - Józsefvárosi Szent Kozma Egészségügyi Központ Tüdőgyógyászat és Gondozó, Budapest
  - Kispesti Egészségügyi Intézet Tüdőgondozó, Ernyőképszűrő állomás, Budapest
  - Szent Kristóf Szakrendelő Tüdőgondozó, Budapest
  - Toldy Ferenc Kórház és Rendelőintézet I. Tüdőgondozó, Cegléd
  - Csornai Margit Kórház Tüdőbeteggondozó Intézet, Csorna
  - Debreceni Egyetem Klinikai Központ, Kenézy Gyula Campus Pulmonológiai részleg, Debrecen
  - Dombóvári Szent Lukács Kórház, Tüdőbeteggondozó, Dombóvár I., Dombóvár
  - Dorogi Szent Borbála Szakkórház és Szakorvosi Rendelő, Dorog
  - Szent Pantaleon Kórház Rendelőintézet Dunaújváros, Dunaújváros
  - Vaszary Kolos Kórház Tüdőgondozó Esztergom, Esztergom
  - Bugát Pál Kórház Tüdőbeteg Gondozó Intézet, Gyöngyös
  - Békés Megyei Központi Kórház 1. Tüdőgyógyászat Szakrendelés, Gyula
  - Jászberényi Szent Erzsébet Kórház Tüdőgyógyászat Járóbeteg ellátás, Jászberény
  - Lumniczer Sándor Kórház-Rendelőintézet Tüdőgondozó, Kapuvár
  - Kátai Gábor Kórház Tüdőgyógyászati Szakrendelés, Karcag
  - Bács-Kiskun Megyei Kórház Tüdőgondozó Szakrendelés, Kecskemét
  - Keszthelyi Kórház Tüdőgondozó, Keszthely
  - Szent Damján Görögkatolikus Kórház Tüdőgyógyászati gondozó 1., Kisvárda
  - Selye János Kórház Tüdőgyógyászati Szakellátás, Komárom
  - Kunszentmárton Városi Egészségügyi Központ Tüdőgyógyászat, Kunszentmárton
  - Szaplonczay Manó Marcali Kórház, Tüdőgyógyászati Szakrendelés, Marcali
  - Mohácsi Kórház, Tüdőbeteggondozó, Mohács
  - Karolina Kórház-Rendelőintézet Mosonmagyaróvár, Mosonmagyaróvár
  - Nagyatádi Kórház Tüdőgondozó, Nagyatád
  - FM Magánklinika Eü. Szolg. Kft., Nyíregyháza
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza
  - Orosházi Kórház Tüdőgondozó, Orosháza
  - Oroszlányi Szakorvosi és Ápolási Intézet Tüdőgyógyászat, Oroszlány
  - Egyesített Egészségügyi Intézmények, Tüdőgondozó, Pécs
  - Szent Lázár Megyei Kórház, Tüdőbeteggondozó Szakrendelő, Salgótarján
  - Sarkadi Kistérségi Egészségügyi Fejlesztő Nonprofit Kft., Sarkad
  - Békés Megyei Képviselő-testület Pándy Kálmán Kórháza Tüdőgondozó, Szeghalom
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintézet Tüdőgyógyászati Szakrendelés, Szolnok
  - Markusovszky Egyetemi Oktatókorház, Szombathely
  - Zala Megyei Szent Rafael Kórház Pulmonológia, Allergológiai és Asztma Szakrendelés, Zalaegerszeg

IPD SHARING:
Plan to Share IPD: No